CLINICAL TRIAL: NCT01132859
Title: VRC 900: Evaluation of Tissue-Specific Immune Responses in Adults 18 Years of Age and Older
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100109; 10-I-0109
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01-09

CONDITIONS: Immunity, Mucosal; Immune System Processes; Blood Specimen Collection
Keywords: Specimen Collection; Mucosal Immunity; Immune Responses; Immunity; Vaccines; Natural History; Healthy Volunteer; HV

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants 18 years of age or older willing to donate blood and tissue specimens and participate in imaging studies to evaluate the components of the immune system

SUMMARY:
Background:

- The Vaccine Research Center (VRC) is dedicated to understanding immune responses associated with prevention and treatment of infectious diseases. To study these immune responses, researchers need to collect specimens and images from individuals who have recently had a vaccination or recovered from an infection. These specimens and images are used to study different diseases and immune responses, and can be used to investigate ways to prevent or treat different medical conditions.

Objectives:

- To evaluate blood and other tissue samples for immune responses to vaccines and natural infections.

Eligibility:

- Healthy volunteers at least 18 years of age who agree to donate specimens for research purposes.

Design:

* Participants will have clinical evaluations and will be asked to provide some of the following samples, depending on the research question being addressed. All procedures and sample donations are optional and voluntary:
* Blood samples through regular blood draws (for whole blood) and apheresis (to collect specific parts of the blood such as plasma or white blood cells)
* Urine, semen, saliva, or vaginal swab samples
* Tissue samples or biopsy specimens
* Undergo procedures such as bronchoscopy (lung and respiratory tract), gastrointestinal endoscopy (stomach and upper intestinal tract), or colonoscopy (lower intestinal tract) to obtain tissue samples
* Undergo imaging studies such as positron emission tomography (PET) or computed tomography (CT) scans

Duration of participation is variable depending on the research question but will usually last up to 1 year.

- Participants will be compensated for participation.

DETAILED DESCRIPTION:
Protocol Design:

This is a specimen and data collection protocol designed with the research purpose of understanding the immune responses to vaccines and infections in adult participants. The information gained will enhance the knowledge of immune correlates of protection and will help in laboratory work related to the development and validation of immunological assays. This protocol will allow Vaccine Research Center (VRC) investigators and collaborators to evaluate tissue level immune responses in participants who are recipients of Food and Drug Administration (FDA)-licensed vaccines, recipients of investigational vaccines, control subjects, and participants naturally infected with infectious diseases as examples of naturally acquired immunity. Immune responses will be evaluated using collection of blood, body fluids, mucosal and tissue samples to perform clinical evaluations for research rather than therapeutic goals. Imaging using ultrasonography may be employed to image tissues such as lymph nodes to guide sampling. Detailed studies of immune responses in blood, body fluids and a diversity of tissue types, including a variety of mucosal surfaces, will further the understanding of immune responses following vaccination or recovery from an infectious disease and will advance development of vaccines against existing, new, and re-emerging pathogens.

Subjects:

Up to 500 participants 18 years of age and older who agree to collection, use, and storage of specimens and images for research purposes will be enrolled. Participants must not be pregnant or breast-feeding for certain study sample collection procedures or to receive FDA-licensed live virus vaccines.

Study Plan:

Participants will receive information about study procedures and, if willing to participate, will sign the study informed consent. FDA-licensed vaccines may be administered to some study participants as part of study participation. As per NIH Clinical Center (CC) policy, where appropriate, participants will provide additional informed consent for study procedures.

Duration:

Individual participants may donate samples as often as permitted by the protocol and NIH CC guidelines. The CC guidance on the volume of blood drawn and other inpatient/outpatient procedures will be followed. The protocol will undergo continuing review by the Institutional Review Board (IRB) annually.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18 years of age or older.
  2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
  3. Able and willing to complete the informed consent process.
  4. Willing to donate specimens for storage to be used for research.

EXCLUSION CRITERIA:

1. Any medical, psychiatric, occupational condition or other condition that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a participant s ability to give informed consent.
2. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), use of anticoagulant medications for an ongoing medical condition, significant bruising or bleeding difficulties with intramuscular injections or blood draws. [Note: Participants taking anticoagulants, such as aspirin, prophylactically may be considered on a case to case basis.]

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants 18 years of age or older willing to donate blood and tissue specimens and participate in imaging studies to evaluate the components of the immune system.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-05-18 (Actual)

PRIMARY OUTCOMES:
To use specimens and accumulated data for enhancement of understanding the correlates of immune protection. | Throughout the study
  By sample collection and imaging studies
To evaluate blood, body fluid, and tissue immune responses and pathogen dynamics of naturally infected and antigen-na(SqrRoot) ve subjects | Throughout the study
  By sample collection and imaging studies
To evaluate innate, humoral, and cellular immune responses and pathogen dynamics in the context of vaccination in the blood, body fluids, excretions, and tissues | Throughout the study
  By sample collection and imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: Lesia K Dropulic, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Querec TD, Akondy RS, Lee EK, Cao W, Nakaya HI, Teuwen D, Pirani A, Gernert K, Deng J, Marzolf B, Kennedy K, Wu H, Bennouna S, Oluoch H, Miller J, Vencio RZ, Mulligan M, Aderem A, Ahmed R, Pulendran B. Systems biology approach predicts immunogenicity of the yellow fever vaccine in humans. Nat Immunol. 2009 Jan;10(1):116-125. doi: 10.1038/ni.1688. Epub 2008 Nov 23. PMID 19029902
- [Background] Wrammert J, Miller J, Akondy R, Ahmed R. Human immune memory to yellow fever and smallpox vaccination. J Clin Immunol. 2009 Mar;29(2):151-7. doi: 10.1007/s10875-008-9267-3. Epub 2008 Dec 4. PMID 19052852
- [Background] Plotkin SA. Vaccines: the fourth century. Clin Vaccine Immunol. 2009 Dec;16(12):1709-19. doi: 10.1128/CVI.00290-09. Epub 2009 Sep 30. PMID 19793898
- [Derived] Herrin DM, Coates EE, Costner PJ, Kemp TJ, Nason MC, Saharia KK, Pan Y, Sarwar UN, Holman L, Yamshchikov G, Koup RA, Pang YY, Seder RA, Schiller JT, Graham BS, Pinto LA, Ledgerwood JE. Comparison of adaptive and innate immune responses induced by licensed vaccines for Human Papillomavirus. Hum Vaccin Immunother. 2014;10(12):3446-54. doi: 10.4161/hv.34408. PMID 25483691
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-I-0109.html